CLINICAL TRIAL: NCT05753332
Title: Association Between Short-term PM2.5 Exposures and Nrf2 Dependent Ferroptosis Pathway
Brief Title: Association Between PM2.5 and Ferroptosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Northern Jiangsu People's Hospital (Other)
Collaborators: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, WenJing Zhao, M.D.; attending doctor, Northern Jiangsu People's Hospital
Other Study IDs: NorthernJiangsu-zhao
Record Dates: First submitted 2023-02-06; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Exposure to Polluted Air
Keywords: PM2.5; Nrf2; Cognitive function; Ferroptosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — the enrolled participant's peripheral whole blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The control group: the invited volunteers live in Yangzhou, Jiangsu, China (low PM2.5 level based on previous official PM2.5 records)
- The PM2.5 exposure group: the invited volunteers live in Xuzhou, Jiangsu, China (high PM2.5 level based on previous official PM2.5 records)

SUMMARY:
This cohort study aims to discover the possible effects of PM2.5 exposures on the Nrf2- dependent ferroptosis pathway. This observational cohort's main question is whether PM2.5 exposures will affect the Nrf2- dependent ferroptosis pathway.

Participants will be divided into two groups: the control group and the air pollution to detect the biomarkers of the Nrf2- dependent ferroptosis pathway.

DETAILED DESCRIPTION:
Background: Despite the exact mechanism of the effects of air pollution (PM2.5) on the central nervous system is still under debate, there is increasing evidence that air pollution (PM2.5) will cause cognitive decline. It is well known that air pollution (PM2.5) will cause the release of proinflammatory cytokines by microglia and cognitive decline. TNF-α plays a key role in cognitive function and our previous research indicated that Nrf2 plays a crucial role in seizures-induced cognitive function (NCT05269901) . However, whether PM2.5-induced TNF-α will further trigger Nrf2- dependent ferroptosis to facilitate cognitive decline is still unexplored. This pilot clinical trial aims to discover the possible association between PM2.5 exposures and the changes in TNF-α level and Nrf2- dependent ferroptosis pathway.

Methods:

1. The investigators first analyze the genes expression of the GSE60767 from the GEO database (www.ncbi.nlm.nih.gov/geo) using the GPL6947 platform
2. The investigators enrolled 30 people and aged-matched PM2.5 exposures people from two cities (Yangzhou and Xuzhou) as the control and air pollution group based on previous PM2.5 records;
3. Recorded the PM2.5 level in two cities every 5 days between 2022.12 and 2023.2 (winter) to compare the difference;
4. TNF-α ELISA KIT was used to compare the proinflammatory cytokines in two groups
5. 4HNE (4-Hydroxynonenal )ELISA KIT was used to compare the lipid reactive oxygen species level in two groups
6. Quantitative reverse transcription PCR (Polymerase Chain Reaction) was used to compare messenger ribonucleic acid (mRNA) expression of the Nrf2-dependent ferroptosis pathway (Nrf2, SLC7A11, GPX4) Detailed Methods protocol

1. PM2.5 level source: the PM2.5 levels were recorded via the data from the Ministry of Ecology and Environment of the People's Republic of China (air.cnemc.cn:18007) 2. The criteria of enrolled participants were as follows：Inclusion: living in this city for more than 3 years; no exposure to any chemistry pollution before; Exclusion: significant changes in biomarkers (TNF-α, Nrf2, SLC7A11, GPX4) at the beginning; neurological disorders; endocrine diseases; cancer 3. Sample collection: At the beginning and the end of this study, the enrolled participant will come to the hospital to collect peripheral Blood (Northern Jiangsu and Xuzhou center, respectively), and the blood samples will be collected into EDTA (ethyleneDiamine tetraacetic acid) vacutainer tubes and then divided into leukocytes and plasma for further experiments 4. TNF-α ELISA KIT: Plasma TNF-α concentrations were detected by the competitive ELISA method 5. 4HNE（4-Hydroxynonenal ）ELISA KIT : Plasma 4HNE concentrations were detected by the competitive ELISA method 6. primer sequence: h-GPX4 forward: 5'-GAGGCAAGACCGAAGTAAACTAC-3' h-GPX4 reverse: 5'-CCGAACTGGTTACACGGGAA-3' h-SLC7A11 forward: 5'-TCTCCAAAGGAGGTTACCTGC-3' h-SLC7A11 reverse: 5'-AGACTCCCCTCAGTAAAGTGAC-3' h-Nrf2 forward 5'-ATAGCTGAGCCCAGTATC-3' h-Nrf2 reverse 5'- CATGCACGTGAGTGCTCT-3' h-GAPDH forward: 5'-GGAGCGAGATCCCTCCAAAAT-3' h-GAPDH reverse: 5'-GGCTGTTGTCATACTTCTCATGG-3'

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years old living in this city for more than one year no exposure to any chemistry pollution before

Exclusion Criteria:

* Aged below 18 years old neurological disorders; endocrine diseases; cancer significant changes in biomarkers (TNF-α, Nrf2, SLC7A11, GPX4) at the beginning

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The control group will be selected from the invited volunteers who live in Yangzhou city via the website, email, and poster.
  The PM2.5 group will be selected from the invited volunteers who live in Xuzhou city via the website, email, and poster.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-02-25 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
4HNE level | From the date of all participants documented baseline data, until the date of the last participant documented the changes of biomarkers in peripheral blood, assessed up to 120 days
  Biomarkers of ferroptosis, an indicator of lipid reactive oxygen species
TNF-α ELISA KIT | From the date of all participants documented baseline data, until the date of the last participant documented the changes of biomarkers in peripheral blood, assessed up to 120 days
  Biomarkers of the proinflammatory cytokines
mRNA expression of the Nrf2- dependent ferroptosis | From the date of all participants documented baseline data, until the date of the last participant documented the changes of biomarkers in peripheral blood, assessed up to 120 days
  Biomarkers of the Nrf2- dependent ferroptosis

CONTACTS AND LOCATIONS:
Overall Officials: Ju Gao, Phd, Study Director — Affiliated Northern Jiangsu People's Hospital of Yangzhou University
Locations (1):
- Wenjing Zhao, Yangzhou, Jiangsu, China